CLINICAL TRIAL: NCT06822881
Title: A Clinical Study to Investigate the Safety, Efficacy, and Cellular Metabolism of CT1190B CAR-T Cell Therapy, in Patients With Moderate to Severe Refractory Systemic Lupus Erythematosus (SLE) or Refractory/Progressive Systemic Sclerosis (SSc)
Brief Title: CT1190B in the Treatment of Patients With Moderate to Severe Refractory Systemic Lupus Erythematosus (SLE) or Refractory/Progressive Systemic Sclerosis (SSc)
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Beijing GoBroad Hospital (Other)
Collaborators: CARsgen Therapeutics Co., Ltd. (Industry)
Responsible Party: Principal Investigator, Jing Pan, Principal Investigator, Beijing GoBroad Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CT1190B-CG11002_03
Record Dates: First submitted 2025-02-07; First posted 2025-02-12 (Actual); Last update posted 2025-09-17 (Actual); Status verified 2025-02

CONDITIONS: Systemic Lupus Erythematosus (SLE); Systemic Sclerosis (SSc)
Keywords: CT1190B
MeSH Terms: conditions — Lupus Erythematosus, Systemic; Scleroderma, Systemic | interventions — Immunotherapy, Adoptive

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- CT1190B CAR-T cells Injection (Experimental): CT1190B cells infusion
  Interventions: Drug: CAR-T Therapy

INTERVENTIONS:
Drug: CAR-T Therapy — CT1190B cells infusion

SUMMARY:
A Clinical Study Exploring CT1190B in the treatment of patients with moderate to severe refractory systemic lupus erythematosus (SLE) or refractory/progressive systemic sclerosis (SSc)

DETAILED DESCRIPTION:
A Clinical Study to Investigate the Safety, Efficacy, and Cellular Metabolism of CT1190B CAR-T Cell Therapy in Patients With moderate to severe refractory systemic lupus erythematosus (SLE) or refractory/progressive systemic sclerosis (SSc)

ELIGIBILITY:
Inclusion Criteria:

1. Voluntary signing of the Informed Consent Form (ICF)
2. Age range: At the time of signing the ICF, the age is between 18 and 60 years old (including 18 and 60 years old), regardless of gender.
3. No systemic active infection within 2 weeks before screening.
4. Contraceptive requirements for participants with child - bearing potential.
5. Negative pregnancy test for women with child - bearing potential. Inclusion Criteria for SLE

<!-- -->

1. Meet the EULAR/ACR 2019 SLE classification criteria with a disease history ≥ 6 months.
2. Treatment and disease activity requirements:

   o Before screening, the participant must have received treatment with glucocorticoids combined with immunosuppressive agents (including cyclophosphamide, mycophenolate mofetil, tacrolimus, methotrexate, cyclosporine, leflunomide) and/or biological agents for ≥ 3 months, with a stable dose for ≥ 2 weeks, and the disease is still in an active state. Oral corticosteroid requirements at the time of screening:

   o If treated with corticosteroids alone, prednisone (or equivalent drug) ≥ 7.5 mg/day.

   o When used in combination with immunosuppressive agents and/or biological agents, there is no minimum daily dose requirement for corticosteroids.
3. Positive antibody test at screening: Positive antinuclear antibody, and/or positive anti-ds-DNA antibody, and/or positive anti-Smith antibody.
4. Disease activity score or organ damage: At the screening stage, the SLEDAI - 2K score is ≥ 7 points
5. Active organ involvement at screening: isolated skin and mucous membrane involvement is not eligible for inclusion.
6. Adequate organ function:

   o Renal function: Defined as a calculated creatinine clearance rate (Cockcroft - Gault) ≥ 50 mL/min without the need for hydration assistance.

   o Bone marrow function: Defined as absolute neutrophil count (ANC) ≥ 1.0×10⁹/L and hemoglobin (Hb) ≥ 60 g/L. Blood transfusion and growth factors should not be used to meet these requirements within 7 days before the inclusion and exclusion screening.

   o Liver function: Defined as alanine aminotransferase (ALT) and aspartate aminotransferase (AST) ≤ 2× the upper limit of normal (ULN), and total bilirubin ≤ 2× the upper limit of normal (ULN).

   o Coagulation function: Defined as international normalized ratio (INR) or activated partial thromboplastin time (APTT) ≤ 1.5×ULN.

   o Lung function: Oxygen saturation (SpO₂) ≥ 92% (measured by pulse oximeter) in room air.
   * Cardiac function: Defined as a left ventricular ejection fraction (LVEF) ≥ 40% as evaluated by echocardiogram (ECHO) within 8 weeks before screening.

Inclusion Criteria for SSc

1. Meet the 2013 EULAR/ACR classification criteria for systemic sclerosis and the diffuse - type manifestation simultaneously.
2. Combined with interstitial pneumonia caused by SSc.
3. Meet the definition of refractory or progressive disease:

   o Refractory disease definition: Ineffective after more than 6 months of conventional treatment, or disease recurrence after remission. Conventional treatment is defined as the use of glucocorticoids (more than 1 mg/kg/d) or cyclophosphamide, and one or more of the following immunomodulatory drugs: antimalarials, azathioprine, mycophenolate mofetil, methotrexate, leflunomide, tacrolimus, cyclosporine, and biological agents including Actemra, Rituxan, belimumab, tabitacicept, etc.
   * Progressive disease definition (in the past 6 months):
   * Skin progression: An increase in mRSS > 10%.
   * Lung disease progression: A 10% decrease in FVC, or a 5% decrease in FVC accompanied by a 15% decrease in DLCO.
4. Important organ function:

   o Renal function: Defined as a calculated creatinine clearance rate (Cockcroft - Gault) ≥ 50 mL/min without the need for hydration assistance.

   o Bone marrow function: Defined as absolute neutrophil count (ANC) ≥ 1.0×10⁹/L and hemoglobin (Hb) ≥ 90 g/L. Blood transfusion and growth factors should not be used to meet these requirements within 7 days before the inclusion and exclusion screening.

   o Liver function: Alanine aminotransferase (ALT) and aspartate aminotransferase (AST) ≤ 2× the upper limit of normal (ULN), and total bilirubin ≤ 2× the upper limit of normal (ULN).

   o Coagulation function: INR ≤ 1.5×ULN, prothrombin time (PT) ≤ 1.5×ULN.

   o Cardiac function: Good hemodynamic stability, left ventricular ejection fraction (LVEF) ≥ 40%.

Exclusion Criteria:

1. Previous history of CAR-T cell or other genetically modified T-cell therapies, or previous major organ transplantation.
2. Use of B-cell targeted drugs (such as rituximab) within 2 months before screening.
3. Allergy or intolerance to lymphodepletion drugs, tocilizumab, or life-threatening allergic reactions, hypersensitivity reactions, or intolerance to the CT1190B preparation or its excipients, or a history of other severe allergies such as anaphylactic shock.
4. Use of corticosteroids ≥ 10 mg/day of prednisone (or equivalent drug) within 10 days before the infusion of CT1190B.
5. Use of immunosuppressive agents that affect T-cells (mycophenolate mofetil, methotrexate, cyclosporine, azathioprine, leflunomide, tacrolimus) within 10 days before the infusion of CT1190B.
6. Use of JAK inhibitors (tofacitinib, baricitinib tablets, ruxolitinib, etc.) within 3 days before the infusion of CT1190B.
7. Vaccination with live-attenuated vaccines, inactivated vaccines, or RNA vaccines within 1 month before screening.
8. Diagnosis of cancer within 2 years before signing the ICF. Exceptions include non-melanoma skin cancer treated by radical therapy, local prostate cancer, biopsy-proven cervical carcinoma in situ or squamous intraepithelial lesions detected by cervical smear, and completely resected breast carcinoma in situ.
9. Undergoing major surgery within 4 weeks before signing the ICF, or planning to undergo major surgery during the study, and the investigator deems it will pose an unacceptable risk to the participant.
10. Positive test for HIV, syphilis, active hepatitis B virus infection, or active hepatitis C virus infection at screening.
11. History of central nervous system diseases before screening, including but not limited to cerebrovascular accident, encephalitis, epilepsy, convulsions/seizures, stroke, severe brain injury, dementia, Parkinson's disease, cerebellar diseases, central nervous system vasculitis, cognitive impairment, organic brain syndrome, or mental illness.
12. History of any of the following cardiovascular diseases within 1 month before screening: Heart failure of class III or IV as defined by the New York Heart Association (NYHA), myocardial infarction, unstable angina, uncontrolled or symptomatic atrial arrhythmia, any ventricular arrhythmia, or other heart diseases of significant clinical significance.
13. Participation in other clinical studies within 3 months before screening or still within five half-lives after the last dose of the drug.
14. Current presence of any uncontrolled active infection, including but not limited to active tuberculosis, etc.
15. History or evidence of suicidal thoughts within 6 months before signing the ICF, or any suicidal behavior within the previous 12 months, and the investigator deems there is a significant suicide risk.
16. Pregnant or breastfeeding women.
17. Poor compliance judged by the investigator, inability or unwillingness to comply with the requirements of the study protocol, or other reasons that make the participant unsuitable for this clinical study.

Exclusion Criteria for SLE

1. Severe lupus nephritis within 2 months before screening, requiring hemodialysis, or receiving prednisone ≥ 100 mg/d or equivalent corticosteroid treatment for ≥ 14 days.
2. Lupus crisis within 1 month before screening, and the investigator deems it inappropriate for the participant to participate in this study.
3. Central nervous system manifestations caused by lupus before screening, including but not limited to lupus headache, seizures, cognitive impairment, impaired intellectual function, visual impairment, etc.
4. History of ≥ grade 2 bleeding within 30 days before screening.
5. Plasmapheresis, plasma separation, or hemodialysis within 14 days before screening.

Exclusion Criteria for SSc

1. FVC ≤ 30% of the predicted value or DLCO (corrected for hemoglobin) ≤ 30% of the predicted value.

2. Combined with severe kidney disease or signs of renal crisis in the participant.

3. Risk of active tuberculosis at screening.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 27 (Estimated)
Dates: Start 2025-02-20 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
The incidence rate and severity of dose limiting toxicity (DLT), adverse events (AE), serious adverse events (SAE), and AESI (adverse events of particular concern) | Within 28 days after infusion for DLT, within 180 days after infusion for AE/SAE, within 12 months after infusion for AESI

SECONDARY OUTCOMES:
Proportion of patients who reach lupus low disease activity status (LLDAS) 6 months after infusion | Six months
Changes in American College of Rheumatology Composite Response Index in Systemic Sclerosis (ACR-CRISS) compared to baseline after 3 months of infusion | 3 months after infusion

CONTACTS AND LOCATIONS:
Locations (1):
- Beijing GoBroad Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No